CLINICAL TRIAL: NCT06200038
Title: Effects of Upper Thoracic Mulligan Mobilization for Pain, Range of Motion and Function in Patients With Mechanical Neck Pain
Brief Title: Effect of Manual Therapy on Non Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-FTR-ÖOP-07
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
Keywords: Mechanical Neck Pain; Thoracic Mobilization; Mulligan; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants did not know the difference between sham and true mobilisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan group (MG) (Experimental): Individuals underwent 11 sessions (every day for the first week, every other day for the next two weeks).Hot pack was applied to the neck and upper trapezius area for 20 minutes.2 channels and 4 electrodes in the neck area; Conventional transcutaneous electrical nerve stimulation (TENS) was applied to the patient for 20 minutes with current transition time: 50-100 microseconds, frequency: 60-120 Hz and mild tingling without causing discomfort.US application was performed at a frequency of 1.5 W/cm2 and 1 Mhz for 8 minutes.Stretching exercises were applied to the trapezius upper part and levator scapula muscles for 15-30 seconds with 10 repetitions under the supervision of a physiotherapist.In addition to physiotherapy applications in MG, Mulligan natural apophyseal reversal technique was applied to the upper thoracic segments. Mulligan mobilization was performed with 3 sets of 10 repetitions and 15-20 seconds of rest between sets.
  Interventions: Other: Mulligan Reverse Natural Apophysial Glide Technique (RNAGS)
- Sham (different in the direction and amplitude of mobilization) group (Sham Comparator): Individuals underwent 11 sessions (every day for the first week, every other day for the next two weeks).Hot pack was applied to the neck and upper trapezius area for 20 minutes.2 channels and 4 electrodes in the neck area; Conventional TENS was applied to the patient for 20 minutes with current transition time: 50-100 microseconds, frequency: 60-120 Hz and mild tingling without causing discomfort.US application was performed at a frequency of 1.5 W/cm2 and 1 Mhz for 8 minutes.Stretching exercises were applied to the trapezius upper part and levator scapula muscles for 15-30 seconds with 10 repetitions under the supervision of a physiotherapist.Sham mobilization was applied to the segments where Mulligan mobilization was carried out in Sham group, in which the direction of thrust and thrust were different.
  Interventions: Other: Conventional physical therapy and sham manual therapy
- Physiotherapy group (Other): Individuals underwent 11 sessions (every day for the first week, every other day for the next two weeks).Hot pack was applied to the neck and upper trapezius area for 20 minutes.2 channels and 4 electrodes in the neck area; Conventional TENS was applied to the patient for 20 minutes with current transition time: 50-100 microseconds, frequency: 60-120 Hz and mild tingling without causing discomfort.US application was performed at a frequency of 1.5 W/cm2 and 1 Mhz for 8 minutes.Stretching exercises were applied to the trapezius upper part and levator scapula muscles for 15-30 seconds with 10 repetitions under the supervision of a physiotherapist.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Mulligan Reverse Natural Apophysial Glide Technique (RNAGS) — Mulligan mobilization techniques was applied to the upper thoracic segments with the RNAGS technique. The application was performed with one hand (thumb in extension, other fingers flexed) that was used to perform the pushing maneuver on the transverse processes, while the other arm was used to gently grasp the head of the patient and recline the neck against the body for stabilization.
  Conventional TENS was applied to the neck area with 2 channels and 4 electrodes for 20 min (current passage time: 50-100 microseconds, frequency: 0-120 Hz). Ultrasonography was performed for 8 minutes with an intensity of 1.5 w/cm2 and a frequency of 1 MHz. Stretching exercises were applied to the upper part of the trapezius and levator scapula muscles for 15-30 seconds for 10 repetitions by a physiotherapist.
  Other Names: TENS; Hotpack; Utrasound; Stretching exercises
  Arms: Mulligan group (MG)
Other: Conventional physical therapy and sham manual therapy — A sham Mulligan RNAGS technique with low pressure compression was applied to thoracic region.
  Conventional TENS was applied to the neck area with 2 channels and 4 electrodes for 20 min (current passage time: 50-100 microseconds, frequency: 0-120 Hz). Ultrasonography was performed for 8 minutes with an intensity of 1.5 w/cm2 and a frequency of 1 MHz. Stretching exercises were applied to the upper part of the trapezius and levator scapula muscles for 15-30 seconds for 10 repetitions by a physiotherapist.
  Other Names: TENS; Hotpack; Utrasound; Stretching exercises
  Arms: Sham (different in the direction and amplitude of mobilization) group
Other: Conventional physical therapy — Conventional TENS was applied to the neck area with 2 channels and 4 electrodes for 20 min (current passage time: 50-100 microseconds, frequency: 0-120 Hz). Ultrasonography was performed for 8 minutes with an intensity of 1.5 w/cm2 and a frequency of 1 MHz. Stretching exercises were applied to the upper part of the trapezius and levator scapula muscles for 15-30 seconds for 10 repetitions by a physiotherapist
  Other Names: TENS; Hotpack; Utrasound; Stretching exercises
  Arms: Physiotherapy group

SUMMARY:
The aim of this study is to investigate the effects of Mulligan concept Reverse Natural Apophysial Glide Technique (RNAGS)technique applied to the thoracic region on pain, limitation of movement, and functionality in individuals with mechanical neck pain.

DETAILED DESCRIPTION:
When we look at the studies investigating the effectiveness of different treatment modalities in non-specific neck pain (NSNP), there is no method accepted as the gold standard for the treatment of NSNP. One of the preferred treatment options for NSNP is physiotherapy and rehabilitation. Physiotherapy and rehabilitation includes electrotherapy modalities, therapeutic exercises, joint mobilisation and manipulations, myofascial release. Among these treatments, manual therapy, which targets the harmony of structure and function, is one of the most preferred treatment methods by physiotherapists. Manual therapy provides improvement by orienting the body's biomechanics, circulation and body structure by directly affecting the joints, muscles and soft tissues. In the literature, there are studies on both cervical mobilisation and thoracic mobilisation for neck pain. Cervical mobilisation and manipulation in neck pain are controversial because they carry certain risks. It has been reported that mobilisation of the thoracic spine decreases pain in the cervical region and increases mobilisation in this region. When the literature was examined, there was no study examining the effect of the Mulligan concept natural apophyseal reversal technique applied to the thoracic region on NSNP. This study was planned to investigate the effect of natural apophyseal reversal on pain and mobility limitation in individuals diagnosed with NSNP.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65
* Those with neck pain lasting at least 3 months
* Individuals diagnosed with mechanical neck pain by a specialist physician

Exclusion Criteria:

* Those with a history of spinal surgery
* Those with a history of whiplash injury
* Those with a history of trauma in the cervical and thoracic region
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Joint Range of Motion Assessment (ROM) | 3 weeks
  Active flexion, extension, right/left lateral flexion and rotation of the cervical region were measured in the sitting position with a phone goniometer application.
Pain Assessment | 3 weeks
  Visual analogue scale (VAS) was used to assess the severity of mechanical neck pain. Individuals were asked to mark the pain they felt on a 10 cm long VAS scale ("0" indicates no pain and "10" indicates unbearable pain).
Neck Disability Status Assessment (NDI) | 3 weeks
  Evaluate neck disability status A questionnaire consisting of 10 items. Seven items are related to activities of daily living, two are related to pain intensity and one is related to concentration. The response to each item is scored between 0 (no limitation) and 5 (maximum limitation) and the final NDI score is obtained by summing each score

CONTACTS AND LOCATIONS:
Overall Officials: Omer Osman PALA, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan for data sharing.